CLINICAL TRIAL: NCT03643042
Title: Impact of 2 Transfusion Strategies on the Quality of Life of Multi-transfused Patients With Low Risk Myelodysplastic Syndrome: Multicenter Randomized Trial Comparing a Liberal vs. Restrictive Transfusion Regimen
Brief Title: Impact of 2 Transfusion Strategies on Quality of Life of Multitransfused Patients With Low-risk Myelodysplastic Syndrome
Acronym: SMD-transfu
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The SMD SEUIL TRANSFU study was stopped prematurely because we encountered enrolment difficulties and new treatments are available on the market for patients with RARS or SFR3B1 mutation (Luspatercept).
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC-P0071
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Myelodysplastic Syndromes; Transfusion-dependent Anemia
Keywords: Myelodysplastic Syndromes; Transfusion; Quality of life; Physical performance
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Blood Transfusion

STUDY DESIGN:
Intervention Model Description: Two modalities of threshold for transfusion:
  * Restrictive group: Hb < 80g/L and Hb maintain between 80 and 100g/L
  * Liberal group: Hb < 100g/L and Hb maintain between 100 and 120g/L
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive group (Experimental): Transfusion with: Hb < 80g/L and Hb maintain between 80 and 100g/L
  Interventions: Other: Transfusion
- Liberal group (Experimental): Transfusion with: Hb < 100g/L and Hb maintain between 100 and 120g/L
  Interventions: Other: Transfusion

INTERVENTIONS:
Other: Transfusion — Transfusion with Hb maintain between 80 and 100g/L or Hb maintain between 100 and 120g/L

SUMMARY:
Myelodysplastic syndromes (MDS) are heterogeneous malignant bone marrow disorders characterized by ineffective haematopoiesis, peripheral blood cytopenias and variable risk of leukaemia transformation.

Anemia is the most common manifestation of bone marrow failure in MDS. After failure with first-line treatment by Erythropoietin, patients survive in average 5 years under long term blood transfusion. Modalities of blood transfusion are not clearly defined.

Then, the objective of this randomized comparative multicentric study is to compare two modalities of threshold for transfusion:

* Restrictive group: Hb < 80g/L and Hb maintain between 80 and 100g/L
* Liberal group: Hb < 100g/L and Hb maintain between 100 and 120g/L

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are heterogeneous malignant bone marrow disorders characterized by ineffective haematopoiesis, peripheral blood cytopenias and variable risk of leukaemia transformation. The median age at diagnosis is 75 years. The incidence is about 30 per 100,000, over 70 years. Etiology is unknown in more than 85% of cases, chemo-induced causes and family cases are well individualized.

Diagnosis, prognosis, and classification (WHO) are based on joint cytologic analysis of peripheral blood, bone marrow, and spinal cytogenetic analysis. The main therapeutic objectives in low-risk MDS are to correct cytopenias, improve quality of life and prevent aggravation of co-morbidities.

Anemia is the most common manifestation of bone marrow failure in MDS. It is encountered in 80% of cases at diagnosis and almost always occurs in the progression of the disease. Its presence and importance have a pejorative prognostic value, but it is not clear whether this anemia is indicative of a more serious clonal disease or whether it is the repercussions of anemia that lead to a more severe prognosis. After failure with first-line treatment by Erythropoietin (EPO), patients survive in average 5 years under long term blood transfusion. Modalities of blood transfusion are not clearly defined.

Studies in the general geriatric population and in cases of acute anemia are in favor of a restrictive transfusion regimen (threshold around 70 g/L), while experience during MDS with EPO suggest that maintaining a higher hemoglobin count could have a favorable impact on quality of life, physical performance, or even survival of patients with MDS.

Then, the objective of this randomized comparative multicentric study is to compare two modalities of threshold for transfusion:

* Restrictive group: Hb < 80g/L and Hb maintain between 80 and 100g/L
* Liberal group: Hb < 100g/L and Hb maintain between 100 and 120g/L

ELIGIBILITY:
Inclusion Criteria:

* Patients with low risk or intermediate risk MDS: Revised International Prognostic Scoring System (IPSS-R) less than or equal to 4.5
* Relapse or failure after Erythropoiesis-Stimulating Agent (ESA) therapy or others treatments (Lenalidomide, Thalidomide, 5-Azacytidine, antithymocyte globulin (ATG), Luspatercept, Decitabine, allograft)
* Transfusion dependent: in average at least 3 transfusion episodes in the last 6 months and total of packed red blood cells (PRBC): more than 8 in the last 12 months and less than 150 in total.
* ≥ 18 years of age
* The Eastern Cooperative Oncology Group (ECOG) score < 4
* Life expectancy > 12 Months
* Patients willing to participate in the study and who have signed the informed consent form

Exclusion Criteria:

* Patients with disease modifying agents for their MDS such as: ESA therapy, Lenalidomide, Thalidomide revlimid, Vidaza, Allograft, antithymocyte globulin (ATG), Luspatercept, Decitabine, experimental agents, other clinical trial, taken within 3 months prior to inclusion (chelators are accepted)
* According to physician: unable to tolerate restrictive or liberal red cell transfusion thresholds (e.g. clinically significant cardio-respiratory failure)
* Cognitive alteration (inability to complete QUALMS)
* Inability to perform the physical performance test Timed up and go test
* Splenomegaly > 3 cm below the costal margin
* Severe renal failure with creatinine clearance < 30ml / min
* Patients presenting with active bleeding or evidence of significant haemolysis
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Quality of Life by Myelodysplasia Scale (QUALMS) score | six months post-randomization
  Quality of Life assessed by a specific validated and adapted disease scale :Quality of Life by Myelodysplasia Scale (QUALMS) score at six months post-randomization. The QUALMS consists of 38 items, and takes less than 10 minutes to complete. Scored on a scale of 0 to 100 higher score is correlated with better MDS-specific quality of life.

SECONDARY OUTCOMES:
Quality of Life by Myelodysplasia Scale (QUALMS) score over the twelve months of follow-up | 3, 6, 12 Months
  Evolution of the QUALMS score over the twelve months of follow-up. Scored on a scale of 0 to 100 higher score is correlated with better MDS-specific quality of life.
Timed up and go test over the twelve months of follow-up | 3, 6, 12 Months
  Evolution of physical performance (the time required for the Timed up and go test) at six months post-randomization and over the twelve months of follow-up
Transfusion incidents rate over the twelve months of follow-up | 3, 6, 12 Months
  Transfusion incidents rate during the twelve months of follow-up among allo-immunization, hospitalization for pulmonary overload, iron overload (ferritin, transferrin saturation), TRALI (Transfusion-Related Acute Lung Injury)
Transfusion costs over the twelve months of follow-up | 3, 6, 12 Months
  Transfusion costs (number of Packed red blood cells (PRBC) used) during the twelve months of follow-up
Time of occurrence of diagnosis of heart and liver damage due to transfusional iron overload over twelve months of follow-up | 3, 6, 12 Months
  Time of occurrence of diagnosis of heart and liver damage due to transfusional iron overload over twelve months of follow-up. The diagnosis will be established according to the standard procedure based on annual MRI, in particular by measuring the LIC (liver iron concentration), the MIC (myocardial iron concentration) and the cardiac T2* value.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pascal, MD, Study Director — GHICL
Locations (19):
- France (19):
  - Abbeville CH, Abbeville
  - Amiens CHU, Amiens
  - Arras CH, Arras
  - Henri Duffaut CH, Avignon
  - Besançon CHU, Besançon
  - Bordeaux CHU, Bordeaux
  - Cote de Nacre CHU, Caen
  - Clermont-Ferrand CHU, Clermont-Ferrand
  - Dunkerque CH, Dunkirk
  - Grenoble CHU, Grenoble
  - Le Mans CH, Le Mans
  - Lens CH, Lens
  - St-Vincent Hospital, Lille
  - Limoges CHRU, Limoges
  - Meaux CH, Meaux
  - Archet 1 Hospital, Nice
  - Saint-Louis Hospital, APHP, Paris
  - Pontchaillou Hospital, Rennes
  - Roubaix CH, Roubaix

IPD SHARING:
Plan to Share IPD: No